CLINICAL TRIAL: NCT06480526
Title: LEGACY (Late Effects of GD2 Antibody and Chemotherapy in Youths): Feasibility of Screening for Early Late Effects of Contemporary Therapy in High-Risk Neuroblastoma Survivors
Brief Title: Feasibility of Screening for Early Late Effects of Contemporary Therapy in High-Risk Neuroblastoma Survivors
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LEGACY; NCI-2024-05183 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-06-14; First posted 2024-06-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: High-risk Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study participant is being asked to be in a research study called LEGACY, because you were treated for high-risk neuroblastoma (HR-NBL).

Primary Objective

To determine the feasibility of conducting comprehensive evaluations, leveraging the established SJLIFE (St. Jude Lifetime Cohort Study) study infrastructure, in survivors of HR-NBL (high-risk neuroblastoma) who are greater than 2 years from completion of contemporary therapy and were previously treated at SJCRH (St. Jude Children's Research Hospital).

Exploratory Objectives

* To describe the health outcomes of survivors of HR-NBL previously treated at SJCRH with contemporary era therapy who are greater than 2 years from completion of therapy.
* To describe the relationship between patient outcomes and social determinants of health (SDOH) in survivors of HR-NBL previously treated at SJCRH with contemporary era therapy who are greater than 2 years from completion of therapy.

DETAILED DESCRIPTION:
The study participant will have blood tests, tests to measure how your nervous system and stomach works, and an ultrasound of your liver for this study. The researchers will test how well your heart and blood vessels are working.

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed with neuroblastoma at < 18 years of age and categorized as high-risk at that time, according to INSS26 or INRGSS27 criteria.
* Participants were treated for HR-NBL at SJCRH on NB2012 or as per NB2012.
* Participants are ≥ 2 years from completion of therapy. Participants are 5 years of age or older.
* Participant or legal guardian is able and willing to give informed consent.
* Participants may choose to participate in all or a fraction of the proposed assessments; refusal to participate in some aspects of the study will not preclude their inclusion.
* Participants must also complete enrollment on SJLIFE.

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Participants who had relapsed or refractory disease during or following completion of modern era treatment for HR-NBL.
* Participants who are pregnant or breastfeeding.
* Participants who are unable to read and understand English

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility will be measured by at least 66% participation rate | Up to 24 months after participant enrollment.
  To determine the feasibility of conducting comprehensive evaluations, leveraging the established SJLIFE (St. Jude Lifetime Cohort Study) study infrastructure, in survivors of HR-NBL (high-risk neuroblastoma) who are greater than 2 years from completion of contemporary therapy and were previously treated at SJCRH (St. Jude Children's Research Hospital). To establish the feasibility, we will estimate the participation rate. The study is considered to have an acceptable participation rate if the 95% lower bound of the participation rate exceeds 66%. Participation is defined as completing ≥ 75% of all proposed assessments.
To describe the health outcomes of survivors of HR-NBL previously treated at SJCRH with contemporary era therapy who are greater than 2 years from completion of therapy. | Health outcomes will be assessed on Days 1, 2, 3, 4, or 5 during the SJLIFE and LEGACY campus visit.
  Participants will go through a comprehensive assessment including the SJLIFE core battery and additional studies in the categories of neurological and autonomic, immunological, quality of life, hematological, renal and metabolic, endocrine, cardiorespiratory, and gastrointestinal (see table below). Their health conditions will be defined by normative data and will be graded using the Revised Common Terminology Criteria for Adverse Events (CTCAE) used by Hudson et al. in SJLIFE studies. The prevalence, cumulative incidence, and latency of selected treatment complications in survivors will be estimated.
  Resting/minimum/maximum heart rate, nerve velocities (median, deep peroneal, common peroneal, Sural), sweat total/baseline/end offset volumes, complete blood cou
Socioeconomic status will be measured by self-reported demographic information | Socioeconomic status, assessed via the household survey, will be assessed on Days 1, 2, 3, 4, or 5 during the LEGACY and SJLIFE campus visit.
  Answers to the household survey, which includes single-item evaluations of self-reported race, ethnicity and primary language, collected per U.S. Health and Human Services guidelines, health literacy utilizing a validated 1-item screen, educational attainment, household materials hardship (HMH), and household income.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Federico, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols